CLINICAL TRIAL: NCT04723147
Title: Dopaminergic Therapy for Inflammation-Related Anhedonia in Depression
Brief Title: DTA (Dopaminergic Therapy for Anhedonia) Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jennifer Felger, Associate Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00000361; 1R61MH121625-01A1 (NIH)
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Depression; Anhedonia
Keywords: Depression; Anhedonia
MeSH Terms: conditions — Depression; Anhedonia | interventions — carbidopa, levodopa drug combination; Levodopa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carbidopa Levodopa followed by Placebo (Experimental): Participants will receive first Carbidopa Levodopa at doses ranging from 150 to 450 mg administered at a ratio of 1 mg carbidopa for every 4 mg L-DOPA with a starting dose of 150 mg/day with dose escalation 150 mg/day per week to a final dose of 450 mg/day; and then placebo.
  Interventions: Drug: Carbidopa Levodopa; Drug: Placebo
- Placebo followed by Carbidopa Levodopa (Experimental): Participants will receive first placebo, and then Carbidopa Levodopa (L-DOPA) at doses ranging from 150 to 450 mg administered at a ratio of 1 mg carbidopa for every 4 mg L-DOPA with a starting dose of 150 mg/day with dose escalation 150 mg/day per week to a final dose of 450 mg/day.
  Interventions: Drug: Carbidopa Levodopa; Drug: Placebo

INTERVENTIONS:
Drug: Carbidopa Levodopa — Patients will receive L-DOPA at doses ranging from 150 to 450 mg administered at a ratio of 1 mg carbidopa for every 4 mg L-DOPA. Starting dose is 150 mg/day with dose escalation 150 mg/day per week to a final dose of 450 mg/day
  Other Names: Sinemet, L-DOPA
Drug: Placebo — A placebo is a sugar pill that has no therapeutic effect and will be administered orally. Participants will receive 1 placebo tablet matching the Carbidopa Levodopa tablet.
  Other Names: Placebo tablet

SUMMARY:
The purpose of this 6-week, double-blind, placebo-controlled, crossover study is to explore new treatment options for people with depression who have high inflammation and anhedonia. Thirty-five male and female participants with depression, between the ages of 25-55 years of age, will be randomized to two study tracks (A and B) to receive both placebo and three doses of L-DOPA, given in different orders. Increases or decreases in each dose will occur gradually over 6 weeks of the study. Participants will complete lab tests, medical and psychiatric assessments, neurocognitive testing and functional MRI (fMRI) scans as part of the study. The total length of participation is about 2 months.

DETAILED DESCRIPTION:
Depression is a widespread disorder (lifetime prevalence >20%). Current antidepressant medications are effective for many patients; however, more than 30% fail to respond. Of the patients that do respond to treatment, some continue to suffer with primary symptoms of depression like an inability to experience pleasure, called anhedonia. In this regard, one biological pathway that may contribute to symptoms of depression and particularly anhedonia is inflammation.

The purpose of this 6-week, double-blind, placebo-controlled, crossover study is to explore new treatment options for people with depression who have high inflammation and anhedonia. Despite evidence of low dopamine function in patients with depression, the ability of existing dopaminergic therapies, like L-DOPA, to affect brain circuits in depression has yet to be explored. This study will help determine the best dose of an FDA-approved medication, Sinemet (L-DOPA) that might be used in the future to treat sub-groups of depressed individuals.

Forty male and female participants with depression, between the ages of 25-55 years of age, will be randomized to two study tracks (A and B) to receive both placebo and three doses of L-DOPA, given in different orders. Increases or decreases in each dose will occur gradually over 6 weeks of the study. Participants will complete lab tests, medical and psychiatric assessments, neurocognitive testing and functional MRI (fMRI) scans as part of the study. The total length of participation is about 2 months.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to give written informed consent;
* men or women, 25-55 years of age
* a primary diagnosis of DSM-V MD, current, as diagnosed by the SCID-I;
* score >10 on the Patient Health Questionnaire [PHQ]-9
* off all antidepressant or other psychotropic therapy (e.g. mood stabilizers, antipsychotics, anxiolytics, and sedative hypnotics) for at least 4 weeks prior to baseline visit (8 weeks for fluoxetine)
* CRP ≥2 mg/L
* Score >/=2 on the anhedonia question of Patient Health Questionnaire [PHQ]-9

Exclusion Criteria:

* history or evidence (clinical or laboratory) of an autoimmune disorder ;
* history or evidence (clinical or laboratory) of hepatitis B or C infection or human immunodeficiency virus infection; - history of any type of cancer requiring treatment with more than minor surgery;
* unstable cardiovascular, endocrinologic, hematologic, hepatic, renal, or neurologic disease (as determined by physical examination, EKG and laboratory testing);
* history of any (non-mood-related) psychotic disorder; active psychotic symptoms of any type; history or current bipolar disorder; history or current gambling disorder; substance abuse/dependence within 6 months of study entry (as determined by SCID);
* active suicidal plan as determined by a score >3 on item #3 on the HAM-D; g. an active eating disorder (except for patients with binge eating disorder in whom binging is clearly associated with worsening of mood symptoms) ;
* a history of a cognitive disorder
* pregnancy or lactation;
* chronic use of non-steroidal anti-inflammatory agents (NSAIDS) (excluding 81mg of aspirin), glucocorticoid containing medications or statins;
* use of NSAIDS, glucocorticoids, or statins at any time during the study;
* urine toxicology screen is positive for drugs of abuse,
* any contraindication for MRI scanning; n. intolerance, sensitivity or contraindication to carbidopa-levodopa (including history of narrow-angle glaucoma, melanoma, gastric and/or duodenal ulcers, bleeding disorders, or frequent migraines).

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Felger, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Only the data - raw and analyzed, or both, depending on the items. Statistical plans an additional information may be shared within the data base but it is not required as the data will be linked to the publications.
Supporting Information: SAP
Time Frame: After publication, within one year of the end of the project.
Access Criteria: Must be NIH investigators and they have to submit an application, including analysis plan, in order to be granted access.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 38 individuals consented to participate in the study and underwent study-specific screening. 19 of these individuals met eligibility criteria and took part in the study. Only those who actually started the study are included in the following tables.
Period: First Intervention
Arm/Group | Carbidopa Levodopa Followed by Placebo | Placebo Followed by Carbidopa Levodopa
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Carbidopa Levodopa Followed by Placebo | Placebo Followed by Carbidopa Levodopa
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carbidopa Levodopa Followed by Placebo | Placebo Followed by Carbidopa Levodopa | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (9.0) | 39.4 (8.6) | 36.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 0 | 2 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Targeted Ventral Striatum to Ventromedial Prefrontal Cortex (VS-vmPFC) Connectivity
Description: Patients will undergo resting-state and task-based functional magnetic resonance imaging (fMRI) to calculate functional connectivity (FC) between the ventral striatum (VS) and ventromedial prefrontal cortex (vmPFC).
  FC is measured as continuous Z scores reflecting the correlation of activity between the brain regions using Fisher's Z transformation {Z(R)=0.5ln[(1+R)/(1-R)]}. This is a standard method for calculating fMRI FC whereby higher FC Z scores reflect stronger connectivity.
Time Frame: Baseline, 1-week of placebo, and 1-week at each dose of L-DOPA (150 mg/day, 300 mg/day and 450 mg/day)
Population: Reported sample sizes reflect the number of available and analyzable fMRI scans for each condition from participants having data at baseline and at least one post L-DOPA or post placebo scan
Measure: Mean (Standard Deviation); unit: Mean subject-level FC Z scores
Groups:
- All Participants: Participants that received Carbidopa Levodopa (150, 300, 450 mg/day per week) and Placebo, independent of the order of administration.
  * Carbidopa Levodopa at doses ranging from 150 to 450 mg administered at a ratio of 1 mg carbidopa for every 4 mg L-DOPA with a starting dose of 150 mg/day with dose escalation 150 mg/day per week to a final dose of 450 mg/day.
  * Placebo: A placebo is a sugar pill that has no therapeutic effect and was administered orally. Participants received 1 placebo tablet matching the Carbidopa Levodopa tablet.
Arm/Group | All Participants
Number analyzed (Participants) | 17
Mean subject-level FC Z scores
  Baseline | 0.183 (0.132)
  Week 1 post- placebo: number analyzed (Participants) | 16
  Week 1 post- placebo | 0.219 (0.125)
  Week 1 post L-DOPA (150 mg/day): number analyzed (Participants) | 15
  Week 1 post L-DOPA (150 mg/day) | 0.275 (0.133)
  Week 1 post L-DOPA (300 mg/day): number analyzed (Participants) | 14
  Week 1 post L-DOPA (300 mg/day) | 0.202 (0.134)
  Week 1 post L-DOPA (450 mg/day): number analyzed (Participants) | 13
  Week 1 post L-DOPA (450 mg/day) | 0.287 (0.135)

2. Secondary Outcome: Effort-Expenditure for Rewards Task (EEfRT)
Description: The EEfRT is a widely used, multi-trial task in which participants are given an opportunity on each trial to choose between two different task difficulty levels in order to obtain monetary rewards. EEfRT will be used as an objective measure of motivation and will be administered following MRI scans during the study. The EEfRT is reported as the percent of high effort trials selected. A higher percentage reflects higher motivation for effort expenditure.
Time Frame: Baseline, 1-week of placebo, and 1-week at each dose of L-DOPA (150 mg/day, 300 mg/day and 450 mg/day)
Population: Reported sample sizes reflect the number of participants with available EEfRT data for each condition.
Measure: Mean (Standard Deviation); unit: percentage of choices
Arm/Group | All Participants
Number analyzed (Participants) | 18
percentage of choices
  Baseline | 0.369 (0.198)
  Week 1 post-placebo: number analyzed (Participants) | 17
  Week 1 post-placebo | 0.300 (0.165)
  Week 1 post L-DOPA (150 mg/day) | 0.368 (0.145)
  Week 1 post L-DOPA (300 mg/day) | 0.322 (0.153)
  Week 1 post L-DOPA (450 mg/day): number analyzed (Participants) | 17
  Week 1 post L-DOPA (450 mg/day) | 0.330 (0.154)

3. Secondary Outcome: Inventory of Depressive Symptomatology- Self-Report (IDS-SR) Anhedonia Scale
Description: Anhedonia symptoms experienced over the past 7 days will be assessed from a subscale of the Inventory of Depressive Symptomatology- Self-Report (IDS-SR), a widely used self-report for measuring depression severity. The anhedonia subscale score is created by summing responses to items #8 (responsiveness of mood to good or desired events), #19 (general interest), and #21 (capacity for pleasure). Total anhedonia subscale scores range from 0-9 with higher scores reflecting greater anhedonia.
Time Frame: Baseline, 1-week of placebo, and 1-week at each dose of L-DOPA (150 mg/day, 300 mg/day and 450 mg/day)
Population: Smaller sample sizes reflect participant withdrawal or incomplete data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 19
score on a scale
  Baseline | 5.2 (2.0)
  Week 1 post-placebo | 3.0 (2.1)
  Week 1 post L-DOPA (150 mg/day): number analyzed (Participants) | 18
  Week 1 post L-DOPA (150 mg/day) | 2.5 (1.5)
  Week 1 post L-DOPA (300 mg/day): number analyzed (Participants) | 18
  Week 1 post L-DOPA (300 mg/day) | 2.4 (1.8)
  Week 1 post L-DOPA (450 mg/day): number analyzed (Participants) | 17
  Week 1 post L-DOPA (450 mg/day) | 3.2 (1.7)

4. Secondary Outcome: Hedonic Capacity as Measured by the Snaith Hamilton Pleasure Clinician Scale (SHAPS-C )
Description: The Snaith-Hamilton Pleasure Scale-Clinician (SHAPS-C) is a clinician-administered version of a validated tool for assessing hedonic tone. The SHAPS-C uses 14 questions. If "Strongly disagree" or "disagree" is chosen as the answer, item receives a score of 1 per question. If "Strongly agree" or "agree" is chosen, item receives a score of 0; then sum the scores. Total possible score ranges from 0 to 14, with higher scores reflecting greater pathology (worse study outcome).
Time Frame: Baseline, 1-week of placebo, and 1-week at each dose of L-DOPA (150 mg/day, 300 mg/day and 450 mg/day)
Population: Smaller sample sizes reflect participant withdrawal or incomplete data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 19
score on a scale
  Baseline | 9.7 (4.1)
  Week 1 post-placebo | 5.6 (5.4)
  Week 1 post L-DOPA (150 mg/day): number analyzed (Participants) | 18
  Week 1 post L-DOPA (150 mg/day) | 3.9 (4.3)
  Week 1 post L-DOPA (300 mg/day): number analyzed (Participants) | 18
  Week 1 post L-DOPA (300 mg/day) | 4.9 (5.1)
  Week 1 post L-DOPA (450 mg/day): number analyzed (Participants) | 18
  Week 1 post L-DOPA (450 mg/day) | 5.3 (5.2)

5. Secondary Outcome: Motivation and Pleasure-Self-Report (MAP-SR)
Description: The Motivation and Pleasure-Self-Report (MAP-SR) will be used to capture self-reported aspects of anhedonia and reduced motivation. The scale uses 18 question each rated on a Likert scale of 0-4. Total possible score ranges from 18 to 72, with higher scores reflecting worse outcome.
Time Frame: Baseline, 1-week of placebo, and 1-week at each dose of L-DOPA (150 mg/day, 300 mg/day and 450 mg/day)
Population: Smaller sample sizes reflect participant withdrawal or incomplete data.
Measure: Mean (Standard Deviation); unit: mean MAP-SR total score
Groups:
- Carbidopa Levodopa (150, 300, 450 mg/Day Per Week) Followed by Placebo: Participants that received Carbidopa Levodopa (150, 300, 450 mg/day per week) and Placebo, independent of the order of administration.
  * Carbidopa Levodopa at doses ranging from 150 to 450 mg administered at a ratio of 1 mg carbidopa for every 4 mg L-DOPA with a starting dose of 150 mg/day with dose escalation 150 mg/day per week to a final dose of 450 mg/day.
  * Placebo: A placebo is a sugar pill that has no therapeutic effect and was administered orally. Participants received 1 placebo tablet matching the Carbidopa Levodopa tablet.
Arm/Group | Carbidopa Levodopa (150, 300, 450 mg/Day Per Week) Followed by Placebo
Number analyzed (Participants) | 19
mean MAP-SR total score
  Baseline | 22.4 (9.9)
  Week 1 post-placebo: number analyzed (Participants) | 18
  Week 1 post-placebo | 35.0 (13.4)
  Week 1 post L-DOPA (150 mg/day): number analyzed (Participants) | 18
  Week 1 post L-DOPA (150 mg/day) | 35.4 (7.0)
  Week 1 post L-DOPA (300 mg/day): number analyzed (Participants) | 18
  Week 1 post L-DOPA (300 mg/day) | 35.3 (5.2)
  Week 1 post L-DOPA (450 mg/day): number analyzed (Participants) | 17
  Week 1 post L-DOPA (450 mg/day) | 33.5 (8.0)

6. Secondary Outcome: Hamilton Depression Rating Scale (HAM-D) Anhedonia and Motivation Item
Description: The anhedonia and motivation-related item from the clinician administered Hamilton Depression Rating Scale (HAM-D) (item #7: work and activities) will be used to measure anhedonia. This item is rated on a scale of 0-4 with higher scores reflecting worse outcome.
Time Frame: Baseline, 1-week of placebo, and 1-week at each dose of L-DOPA (150 mg/day, 300 mg/day and 450 mg/day)
Population: Lower sample sizes reflect participant withdrawal or incomplete data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Carbidopa Levodopa (150, 300, 450 mg/Day Per Week) Followed by Placebo
Number analyzed (Participants) | 19
score on a scale
  Baseline | 3.0 (0.3)
  Week 1 post-placebo | 1.9 (1.1)
  Week 1 post L-DOPA (150 mg/day): number analyzed (Participants) | 18
  Week 1 post L-DOPA (150 mg/day) | 1.6 (1.1)
  Week 1 post L-DOPA (300 mg/day): number analyzed (Participants) | 18
  Week 1 post L-DOPA (300 mg/day) | 1.3 (0.9)
  Week 1 post L-DOPA (450 mg/day): number analyzed (Participants) | 18
  Week 1 post L-DOPA (450 mg/day) | 1.8 (1.0)

ADVERSE EVENTS:
Time Frame: From time of treatment onset (placebo or carbidopa levodopa) up to 6-weeks post-intervention, about 2 months total
Description: Enrolled participants were monitored closely by study clinicians for any adverse events. If any overt study-related adverse events occur, a decision was made about study continuation. Additionally, a record of adverse events for study participants was reported to the DSMB on a regular basis. Subjects were closely monitored during the course of the study for development of any serious or unexpected adverse reactions.
Groups:
- Carbidopa Levodopa, 150 mg: Patients received L-DOPA at 150 mg dose administered at a ratio of 1 mg carbidopa for every 4 mg L-DOPA.
- Carbidopa Levodopa, 300 mg: Patients received L-DOPA at 300 mg dose administered at a ratio of 1 mg carbidopa for every 4 mg L-DOPA.
- Carbidopa Levodopa 450 mg: Patients received L-DOPA at 450 mg dose administered at a ratio of 1 mg carbidopa for every 4 mg L-DOPA.
- Placebo: Participants received 1 placebo tablet matching the carbidopa Levodopa tablet.
Arm/Group | Carbidopa Levodopa, 150 mg | Carbidopa Levodopa, 300 mg | Carbidopa Levodopa 450 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 12/18 | 11/18 | 11/18 | 5/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carbidopa Levodopa, 150 mg (N=18) | Carbidopa Levodopa, 300 mg (N=18) | Carbidopa Levodopa 450 mg (N=18) | Placebo (N=19)
Mild gas (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mild Blurry vision when adjusting to glasses (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mild foot injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nose bleed (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mild Nausea (Gastrointestinal disorders) | 3 (3) | 3 (5) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 7 (9) | 6 (6) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Irritability (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest tightness (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mild Crawling skin sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Mild bruising of venipuncture (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mild bruising on arm from workplace accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus Congestion (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea and vomiting (Food poisoing) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle pain (soreness) (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Weight loss (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased Appetite (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot Flashes (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemiparesthesia with pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panic Attack during MRI scan (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soar throat (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bleeding hemorroid (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal Congestion (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomach cramp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mild allergic reaction to food (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mild pain under lower rib cage (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT04723147/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT04723147/ICF_000.pdf